CLINICAL TRIAL: NCT03572361
Title: Open Label, One-arm, 3-month Study of Once-daily Tablet of V3-MOMMO as Immunotherapy of Breast Cancer
Brief Title: Open Label Immunotherapy Trial for Breast Cancer
Acronym: V3-MOMMO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immunitor LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V3-MOMMO-01
Record Dates: First submitted 2018-06-16; First posted 2018-06-28 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm, open label Phase II study in volunteers with breast cancer receiving daily dose of one pill of vaccine V3-MOMMO
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V3-MOMMO (Experimental): Oral once daily pill of tableted vaccine (V3-MOMMO) containing pooled breast cancer antigens administered for 3 months in 20 volunteers with breast cancer
  Interventions: Biological: V3-MOMMO

INTERVENTIONS:
Biological: V3-MOMMO — Tableted vaccine (V3-OVA) containing breast cancer antigens administered once daily for 3 months

SUMMARY:
This Phase II will evaluate a new type of breast cancer immunotherapy based on a fundamentally new approach that has been successfully tested in a published clinical study of liver cancer. Investigators will test new tableted preparation, V3-MOMMO, obtained from hydrolyzed, inactivated blood and tumors of patients with breast cancer. Study will last 3 months, 20 patients will be recruited, given one pill per day for three months. The primary clinical endpoint is effect on tumor size and burden after 3 months. Secondary endpoint will be effect on levels of tumor markers on monthly basis compared to baseline.

DETAILED DESCRIPTION:
Worldwide, breast cancer is the number one cancer in women. It affects about 12% or 1.7 mln women worldwide. In Mongolia breast cancer is less common, occupies 5-th place by frequency in women, the incidence is 118 per 100,000 or 1,770 cases per year.

Many different types of immunotherapy (especially checkpoint inhibitors) are being tested, but so far the successes have been insignificant, and serious side effects are frequent and unpredictable. This Phase II will evaluate a new type of breast cancer immunotherapy based on a fundamentally new approach that has been successfully tested in a published clinical study of liver cancer. Investigators will test new tableted preparation, V3-MOMMO, obtained from hydrolyzed, inactivated blood and tumor tissues of patients with breast cancer. Study will last 3 months, 20 patients will be recruited, given one pill per day for three months. The primary clinical endpoint is effect on tumor size and lymph nodes burden after 3 months. Secondary endpoint will be effect on levels of tumor markers (i.e., cancer antigen 15-3 (CA 15-3), cancer antigen 27.29 (CA 27.29), and carcinoembryonic antigen (CEA) on monthly basis compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of breast cancer positive at least for CEA tumor marker at above normal threshold level

Exclusion Criteria:

* Mastectomy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Majority of subjects with breast cancer are females
Enrollment: 20 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect on tumor size | Monthly for 3 months
  Changes in tumor size and lymph node burden (if any) compared to baseline

SECONDARY OUTCOMES:
Effect on level of serum tumor markers compared to baseline | Monthly for three months
  Commonly measured tumor markers associated with breast cancer, primarily CA 15-3, CA 27.29, and CEA, at baseline and at study termination

CONTACTS AND LOCATIONS:
Overall Officials: Aldar Bourinbayar, PhD, MD/PhD, Principal Investigator — Immunitor LLC
Locations (1):
- Immunitor LLC, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tarakanovskaya MG, Chinburen J, Batchuluun P, Munkhzaya C, Purevsuren G, Dandii D, Hulan T, Oyungerel D, Kutsyna GA, Reid AA, Borisova V, Bain AI, Jirathitikal V, Bourinbaiar AS. Open-label Phase II clinical trial in 75 patients with advanced hepatocellular carcinoma receiving daily dose of tableted liver cancer vaccine, hepcortespenlisimut-L. J Hepatocell Carcinoma. 2017 Apr 12;4:59-69. doi: 10.2147/JHC.S122507. eCollection 2017. PMID 28443252